CLINICAL TRIAL: NCT02584439
Title: Effect of Pharmacological Heart Rate Reduction on Visco-elastic Properties of the Arterial Wall (BRADYVASC)
Acronym: BRADYVASC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015/077/HP; 2015-002060-17 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Vascular Stiffness; Aging
Keywords: ivabradine; heart rate; aging; visco-elasticity
MeSH Terms: interventions — Ivabradine; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ivabradine-placebo (Other): Volunteers will receive, at meal, ivabradine 5 mg morning and evening for the first period of treatment during 8 days (1 capsule on day 1 and then 1 capsule 2 times a day from day 2 to day 7 and 1 capsule on day 8). A wash out period (12 to 16 days) will follow this first period of treatment. of wash-out . Then, volunteers will receive, at meal, lactose capsule (placebo) morning and evening for the first period of treatment during 8 days (1 capsule on day 1 and then 1 capsule 2 times a day from day 2 to day 7 and 1 capsule on day 8).
  Interventions: Drug: ivabradine; Drug: lactose capsule (placebo)
- placebo-ivabradine (Other): Volunteers will receive, at meal, lactose capsule (placebo) morning and evening for the first period of treatment during 8 days (1 capsule on day 1 and then 1 capsule 2 times a day from day 2 to day 7 and 1 capsule on day 8). A wash out period (12 to 16 days) will follow this first period of treatment. of wash-out . Then, volunteers will receive, at meal, ivabradine 5 mg morning and evening for the first period of treatment during 8 days (1 capsule on day 1 and then 1 capsule 2 times a day from day 2 to day 7 and 1 capsule on day 8).
  Interventions: Drug: ivabradine; Drug: lactose capsule (placebo)

INTERVENTIONS:
Drug: ivabradine — It is a cross over study with two arms : either ivabradine-placebo or placebo-ivabradine. The capsules containing the placebo or ivabradine are completely identical.
  Other Names: Procoralan
Drug: lactose capsule (placebo) — It is a cross over study with two arms : either ivabradine-placebo or placebo-ivabradine. The capsules containing the placebo or ivabradine are completely identical.

SUMMARY:
The conduit arteries exhibit a viscoelastic behavior. Visco-elasticity is partially regulated by endothelium and contributes to the optimization of the heart-vessel coupling. Aging or high resting heart rate (HR) could alter visco-elastic properties leading to increase stiffness of the conduit arteries, an independent cardiovascular risk factor, and degradation of heart-vessel coupling. Lowering HR with ivabradine could reduce these effects.

The objective of this study is to assess the effect of HR reduction by repeated administration of ivabradine on visco-elastic properties, vascular geometry and function of common carotid artery, and on cardiovascular hemodynamic in healthy subject. The influence of aging on ivabradine effects are studied too.

30 healthy volunteers aged between 25 and 65 years old, with a HR ≥ 70 bpm, will receive ivabradine or placebo during 8 days in a single center, randomized, cross-group, double blinded, placebo-controlled study. Each period of treatment will be separate by 12 to 16 days of wash-out. Each subject will participate in an exploration visit, including evaluation of visco-elastic properties, vascular geometry and function of common carotid artery, and cardiovascular hemodynamic, before and after ivabradine or placebo taking.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Caucasian
* Resting heart rate ≥70 bpm (mean of 3 measures after 15 minutes of rest)
* No significant EKG abnormality
* No significant biological abnormalities at inclusion
* Healthy volunteers able to read and understand information letter and to give written informed consent
* Healthy volunteers with medical insurance
* Contraception for two months for women of childbearing age (Estrogen contraceptive or intrauterine device or tubal ligation) (NB : women with amenorrhea for more than 2 years will be considered postmenopausal)

Exclusion Criteria:

* Subjects who don't understand french language
* Person deprived of liberty by an administrative or judicial decision or protected adult subject (under guardianship)
* Pregnant women, nursing mother or women without contraception
* Healthy volunteers who participate to an other trial / participated to an other trial without drugs during the last month or a trial with drugs during the last 3 months
* Hypersensitivity to the active substance or to any of the excipients
* Congenital galactosemia, lactase deficiency, or glucose-galactose malabsorption
* Body mass index (BMI) < 18 kg/m² or > 30 kg/m²
* Severe hypotension (< 90/50 mmHg) (3 measures after 15 minutes of rest)
* Essential or secondary Hypertension (SBP ≥140 mmHg and/or DBP ≥90 mmHg) (3 measures after 15 minutes of rest)
* Active smoking at the day of inclusion (>5 cigarettes/day)
* Severe hypercholesterolemia (Total cholesterol >2,5 g/L)
* Practice sports intensively (≥ 1 hour/day)
* Renal insufficiency (creatinine clearance ≤ 60 ml/min/1,73 m² Cockroft and Gault formula)
* Known liver failure
* Known heart failure or suspected heart failure (congestive episode)
* Atrial fibrillation
* High-grade conduction block (Sick sinus syndrome, sino-atrial block or grade 2 or 3 atrio-ventricular block)
* Abnormal corrected QT with Bazett formula (cQT > 450 ms (men) or > 470 ms (women)).
* Pacemaker
* All cardiac or extra cardiac diseases, active or with sequelae, which, in the opinion of the investigator, is accompanied by a risk of cardiac or vascular consequences
* Retinal disease
* Taking any medication is prohibited during the study except oral contraceptive, acetaminophene or decision of the investigator. In addition, the administration of drugs listed in schedule 2 during the previous 4 weeks prohibits inclusion.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in viscosity of the common carotid artery | 8 days after first administration of ivabradine or placebo

SECONDARY OUTCOMES:
Change from baseline in diameter of the common carotid artery | 8 days after first administration of ivabradine or placebo
Change from baseline in intima-media thickness of the common carotid artery | 8 days after first administration of ivabradine or placebo
Change from baseline in carotid distensibility | 8 days after first administration of ivabradine or placebo
Change from baseline in carotid-femoral pulse wave velocity | 8 days after first administration of ivabradine or placebo
Change from baseline in plasma levels of biomarkers of endothelial function | 8 days after first administration of ivabradine or placebo
Change from baseline in peripheral and central pressures | 8 days after first administration of ivabradine or placebo
Change from baseline in Buckberg index | 8 days after first administration of ivabradine or placebo
Change from baseline in cardiac output | 8 days after first administration of ivabradine or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Roca, MD, Principal Investigator — University Hospital, Rouen; Robinson Joannides, MD,PhD, Study Chair — University Hospital, Rouen
Locations (1):
- Department of Pharmacology, Rouen university Hospital, Rouen, France

REFERENCES:
- [Background] Franklin SS, Khan SA, Wong ND, Larson MG, Levy D. Is pulse pressure useful in predicting risk for coronary heart Disease? The Framingham heart study. Circulation. 1999 Jul 27;100(4):354-60. doi: 10.1161/01.cir.100.4.354. PMID 10421594
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Benetos A, Rudnichi A, Thomas F, Safar M, Guize L. Influence of heart rate on mortality in a French population: role of age, gender, and blood pressure. Hypertension. 1999 Jan;33(1):44-52. doi: 10.1161/01.hyp.33.1.44. PMID 9931080
- [Background] Lantelme P, Mestre C, Lievre M, Gressard A, Milon H. Heart rate: an important confounder of pulse wave velocity assessment. Hypertension. 2002 Jun;39(6):1083-7. doi: 10.1161/01.hyp.0000019132.41066.95. PMID 12052846
- [Background] Bellien J, Iacob M, Remy-Jouet I, Lucas D, Monteil C, Gutierrez L, Vendeville C, Dreano Y, Mercier A, Thuillez C, Joannides R. Epoxyeicosatrienoic acids contribute with altered nitric oxide and endothelin-1 pathways to conduit artery endothelial dysfunction in essential hypertension. Circulation. 2012 Mar 13;125(10):1266-75. doi: 10.1161/CIRCULATIONAHA.111.070680. PMID 22412088
- [Background] Fox K, Ford I, Steg PG, Tendera M, Ferrari R; BEAUTIFUL Investigators. Ivabradine for patients with stable coronary artery disease and left-ventricular systolic dysfunction (BEAUTIFUL): a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Sep 6;372(9641):807-16. doi: 10.1016/S0140-6736(08)61170-8. Epub 2008 Aug 29. PMID 18757088
- [Background] Bellien J, Remy-Jouet I, Iacob M, Blot E, Mercier A, Lucas D, Dreano Y, Gutierrez L, Donnadieu N, Thuillez C, Joannides R. Impaired role of epoxyeicosatrienoic acids in the regulation of basal conduit artery diameter during essential hypertension. Hypertension. 2012 Dec;60(6):1415-21. doi: 10.1161/HYPERTENSIONAHA.112.201087. Epub 2012 Oct 22. PMID 23090775
- [Background] Reil JC, Tardif JC, Ford I, Lloyd SM, O'Meara E, Komajda M, Borer JS, Tavazzi L, Swedberg K, Bohm M. Selective heart rate reduction with ivabradine unloads the left ventricle in heart failure patients. J Am Coll Cardiol. 2013 Nov 19;62(21):1977-1985. doi: 10.1016/j.jacc.2013.07.027. Epub 2013 Aug 7. PMID 23933545
- [Background] Joannides R, Moore N, Iacob M, Compagnon P, Lerebours G, Menard JF, Thuillez C. Comparative effects of ivabradine, a selective heart rate-lowering agent, and propranolol on systemic and cardiac haemodynamics at rest and during exercise. Br J Clin Pharmacol. 2006 Feb;61(2):127-37. doi: 10.1111/j.1365-2125.2005.02544.x. PMID 16433867
- [Background] Boutouyrie P, Beaussier H, Achouba A, Laurent S; EXPLOR trialists. Destiffening effect of valsartan and atenolol: influence of heart rate and blood pressure. J Hypertens. 2014 Jan;32(1):108-14. doi: 10.1097/HJH.0000000000000014. PMID 24275838
- [Background] Tropeano AI, Boutouyrie P, Pannier B, Joannides R, Balkestein E, Katsahian S, Laloux B, Thuillez C, Struijker-Boudier H, Laurent S. Brachial pressure-independent reduction in carotid stiffness after long-term angiotensin-converting enzyme inhibition in diabetic hypertensives. Hypertension. 2006 Jul;48(1):80-6. doi: 10.1161/01.HYP.0000224283.76347.8c. Epub 2006 May 15. PMID 16702490
- [Background] Fox K, Ford I, Steg PG, Tardif JC, Tendera M, Ferrari R; SIGNIFY Investigators. Ivabradine in stable coronary artery disease without clinical heart failure. N Engl J Med. 2014 Sep 18;371(12):1091-9. doi: 10.1056/NEJMoa1406430. Epub 2014 Aug 31. PMID 25176136
- [Background] Drouin A, Gendron ME, Thorin E, Gillis MA, Mahlberg-Gaudin F, Tardif JC. Chronic heart rate reduction by ivabradine prevents endothelial dysfunction in dyslipidaemic mice. Br J Pharmacol. 2008 Jun;154(4):749-57. doi: 10.1038/bjp.2008.116. Epub 2008 Apr 14. PMID 18414390
- [Background] Williams B, Lacy PS, Thom SM, Cruickshank K, Stanton A, Collier D, Hughes AD, Thurston H, O'Rourke M; CAFE Investigators; Anglo-Scandinavian Cardiac Outcomes Trial Investigators; CAFE Steering Committee and Writing Committee. Differential impact of blood pressure-lowering drugs on central aortic pressure and clinical outcomes: principal results of the Conduit Artery Function Evaluation (CAFE) study. Circulation. 2006 Mar 7;113(9):1213-25. doi: 10.1161/CIRCULATIONAHA.105.595496. Epub 2006 Feb 13. PMID 16476843
- [Background] Bolduc V, Drouin A, Gillis MA, Duquette N, Thorin-Trescases N, Frayne-Robillard I, Des Rosiers C, Tardif JC, Thorin E. Heart rate-associated mechanical stress impairs carotid but not cerebral artery compliance in dyslipidemic atherosclerotic mice. Am J Physiol Heart Circ Physiol. 2011 Nov;301(5):H2081-92. doi: 10.1152/ajpheart.00706.2011. Epub 2011 Sep 16. PMID 21926346
- [Background] Maltete D, Bellien J, Cabrejo L, Iacob M, Proust F, Mihout B, Thuillez C, Guegan-Massardier E, Joannides R. Hypertrophic remodeling and increased arterial stiffness in patients with intracranial aneurysms. Atherosclerosis. 2010 Aug;211(2):486-91. doi: 10.1016/j.atherosclerosis.2010.04.002. Epub 2010 Apr 13. PMID 20452592